CLINICAL TRIAL: NCT02497651
Title: Effect of Smoking on Postprandial Gastric Emptying, Glucose Tolerance and Secretion of Gut and Pancreatic Hormones
Acronym: SmokinGLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: h-1-2013-042
Record Dates: First submitted 2015-06-25; First posted 2015-07-14 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
Keywords: Smoking; Diabetes; Incretin hormones; Glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy, heavy smoking men (Experimental): Twelve healthy, male subjects. Intervention: Will undergo two separate, identical test days. One absent smoking, and one with concomitant smoking.
  Interventions: Dietary Supplement: Liquid mixed meal; Other: Skin Biopsy
- Healthy, non-smoking men (Experimental): Twelve healthy, male subjects. Intervention: Will undergo a liquid mixed meal test and a skin biopsy.
  Interventions: Dietary Supplement: Liquid mixed meal; Other: Skin Biopsy

INTERVENTIONS:
Dietary Supplement: Liquid mixed meal — The subjects will ingest a 400 ml chocolate drink, rich on carbohydrates, fat and lipids. In the following 4 hours, blood samples will be drawn from a PVC for the measurement of plasma glucose, gut- and pancreatic hormones, acetaminophen etc. After the 4 hours, the subjects will be offered an ad libitum meal.
Other: Skin Biopsy — All subjects will undergo a skin biopsy procedure. Two small (3 mm) biopsies will be taken from the hip area under local anaesthesia. Standard wound treatment will follow.

SUMMARY:
The study aims to evaluate the effect of smoking on postprandial responses such as plasma glucose, secretion of gut - and pancreatic hormones and gastric emptying in healthy, heavy smoking men.

DETAILED DESCRIPTION:
Epidemiological studies show that active smoking increases the risk of type 2 diabetes in a dose-dependent fashion. Smokers seem to be characterized by central obesity, increased inflammatory markers and oxidative stress, which may lead to insulin resistance and irregularities in glucose metabolism. The current study is a meal test study, in which the aim is to examine a number of variables during a liquid mixed meal test (including gastric emptying, glucose tolerance, gut and pancreatic hormone responses, gall bladder emptying, appetite and food intake) performed in healthy non-smoking subjects and in healthy smokers with or without concomitant cigarette smoking.

The investigators hypothesize that smoking-induced increases in circulating nicotine levels and simultaneous activation of nicotinic receptors in the gastrointestinal tract and in the autonomic nervous system would have detrimental effect on postprandial glucose metabolism and, thus, constitute an important link between smoking and the risk of type 2 diabetes. The current study will help to clarify this hypothesis and improve our general understanding of the association between smoking and gut hormone secretion, gastric emptying and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Both groups

  * Caucasian ethnicity
  * Healthy males
  * Normal haemoglobin
  * Age above 18 years
  * Informed and written consent
  * BMI >20 kg/m2

Smokers • Minimum 20 cigarettes pr. day for at least 1 year

Non-smokers

• No smoking on a regular basis

Exclusion Criteria:

* Both groups

  * Diabetes or prediabetes (fasting plasma glucose levels >6.5 mM or HbA1c >6.0%)
  * First- or second-degree relatives with diabetes
  * Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
  * Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
  * Hypo- or hyperphosphataemia
  * Nephropathy (serum creatinine >150 µM and/or albuminuria
  * Treatment with medicine that cannot be paused for 12 hours
  * Hypo- or hypercalcaemia
  * Hypo- and hyperthyroidism
  * Treatment with oral anticoagulants
  * Active or recent malignant disease
  * Any treatment or condition requiring acute or sub-acute medical or surgical intervention
  * Any condition considered incompatible with participation by the investigators

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postprandial response of glucagon-like peptide-1 (GLP-1) | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)

SECONDARY OUTCOMES:
Postprandial response of insulin | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Postprandial response of Glukagon | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Postprandial response of CCK | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Postprandial response of Gastrin | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Postprandial response of GIP | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Postprandial increment in plasma glucose | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Blood Inflammatory and metabolic markers (composite) | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min)
Gall bladder volume | -30, 20, 40, 80, 240 minutes (meal tests start at 0 min)
  Assessment of gall bladder volume will be mediated by ultrasound
Gastric emptying | -30, -20, -10, 0, 10, 20, 30, 50, 70, 90, 120, 150, 180, 240 minutes (meal tests start at 0 min
  Measurement of acetaminophen is taken as a measure of gastric emptying
GLP-1 receptor expression in the skin | After the 240 minutes
  Analysis of the skin cells from the biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Department of Medicine, Gentofte Hospital, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Derived] Grondahl MF, Bagger JI, Lund A, Faurschou A, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Effects of Smoking Versus Nonsmoking on Postprandial Glucose Metabolism in Heavy Smokers Compared With Nonsmokers. Diabetes Care. 2018 Jun;41(6):1260-1267. doi: 10.2337/dc17-1818. Epub 2018 Mar 30. PMID 29602793